CLINICAL TRIAL: NCT00935051
Title: Assessment of the MMP-1/TIMP-1 Ratio as a Predictor of Wound Healing in Diabetic Foot Ulcers
Brief Title: Matrix Metalloproteinase-1/Tissue Inhibitor of Metalloproteinase-1 (MMP-1/TIMP-1) Ratio and Diabetic Foot Ulcers
Acronym: DIAB-MMP2
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2008-A00155-50
Record Dates: First submitted 2009-07-02; First posted 2009-07-08 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Diabetic Foot Ulcer
Keywords: type 1 diabetes; type 2 diabetes; Diabetic foot ulcer
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Matrix Metalloproteinases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): There is only one group of patients. Thus there is only one arm. Sample of wound fluid will be collected using a non traumatic procedure at week 0 and week 4. A numeric photograph of the wound will be taken at week 0, week 4 and week 12.
  Interventions: Other: Picture + MMPs and TIMP1 at week 0 and week 4

INTERVENTIONS:
Other: Picture + MMPs and TIMP1 at week 0 and week 4 — Sample of wound fluid will be collected using a non traumatic procedure at week 0 and week 4. This will allow to assess the level of MMP9, MMP13, MMP1 and TIMP1. A numeric photograph of the wound will be taken at week 0, week 4 and week 12 in order to assess wound area.

SUMMARY:
The primary objective of this study is to assess the sensitivity and specificity of a MMP-1/TIMP-1 ratio equal to 0.24 at study entry to predict wound healing at 12 weeks' follow up visit.

DETAILED DESCRIPTION:
This monocentric, prospective, non-randomized study assesses the amount of the main metalloproteinases (MMP1, MMP9, MMP13) and their inhibitor TIMP-1 in wound fluid from diabetic foot ulcers.

It aims at demonstrating whether a MMP-1/TIMP-1 ratio equal to 0.24 at study entry can predict wound healing 12 weeks later. All patients will receive the same treatment according to our local protocol. The difference with standard care will be a sample of wound fluid at week 0 and week 4 and a numeric photograph for wound area measurement at week 0, week 4 and week 12.

The main outcome measurement is the percent change of wound area between week 0 and week 12 Secondary objectives include the evaluation of a MMP-1/TIMP-1 ratio equal to 0.4 and the search for confounding factors. A correlation between MMP-9, MMP-13 and wound healing will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 or type 2 diabetes
* Age over 40
* Chronic diabetic foot ulcer (duration over 30 days)
* Grade 1 to 3, stage A and C according to the University of Texas Wound Classification, except stage B and D
* Wound area over 0.5 cm²
* Social Security membership or benefit from Social Security
* Informed consent, with a signed and approved form
* Possibility to have clinical follow-up and compliance during 3 months

Exclusion Criteria:

* Urgent need for locoregional surgery
* Clinical criteria for infection, defined by the presence of pus or/and at least 2 local signs among the following: heat, erythema, lymphangitis, lymphadenopathy, oedema, pain
* Other pathology that could interfere with the healing process (vasculitis, connectivitis, dysimmunity, immunosuppressive treatment or corticoids, ongoing radiotherapy or chemotherapy )
* Any severe pathology that would constitute a contra-indication to the patient's inclusion
* Ongoing therapeutic research protocol
* Underage patient, major patient under guardianship or protected by the Law
* Pregnant, parturient or breastfeeding woman
* Person with no freedom (prisoner), person in an emergency situation, person hospitalized without consent and not protected by the Law

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2009-05; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
MMP-1/TIMP-1 ratio at Week 0 assessed by ELISA and percent change in wound area of diabetic foot ulcer between week 0, week 4 and week 12 | Week 0, week 4 and week 12

SECONDARY OUTCOMES:
Evaluation of a MMP-1/TIMP-1 ratio = 0.4 at Week 0 as a predictor of wound healing at week 12 | Week 0, week 4 and week 12
Recognized clinical prognostic factors such as wound duration, wound area, wound depth and other possible confounding factors affecting the validity of the MMP-1/TIMP-1 ratio | Week 0 to Week 12
Correlation between MMP9, MMP13, MMP9/TIMP1 and MMP13/ TIMP1 ratios and wound healing expressed by the percent change in wound area between week 0, week 4 and week 12. | Week 0 and week 4

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves Benhamou, PhD, Study Director — University Hospital, Grenoble
Locations (2):
- France (2):
  - Diabetology department, Grenoble, Isere
  - Service de Diabétologie du Pr Halimi, CHU Grenoble, Grenoble